CLINICAL TRIAL: NCT01042327
Title: Study to Assess Clearances and Bio-compatibility of ELISIO Dialyzer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Royal Free Hampstead NHS Trust (Other)
Responsible Party: A Davenport, Center for nephrology, University College London Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08/H0724/11
Record Dates: First submitted 2010-01-04; First posted 2010-01-05 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2009-02

CONDITIONS: Chronic Kidney Disease
Keywords: solute clearances
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- dialyzer comparison (Experimental): Stable chronic kidney dialysis patients, currently dialyzing on the main Royal Free hospital dialysis unit will be asked to participate in the study. It is aimed to recruit 15 patients currently dialysing using the Fresenius FX100 dialyzer, who have used Fresenius polysulphone membranes for > 3 months.
  During a mid week dialysis session, dialysis adequacy will be assessed by on line clearance, and samples of both blood and dialysate taken to assess, both clearances and bio-compatibility.
  Thereafter patients would be switched to dialyse using the ELISIOTM-H dialyzer, but continue with the same dialysis prescription, and after 3 months, measurements repeated
  Interventions: Device: ELISIO dialyzer; Device: Fresenius FX100 dialyzer

INTERVENTIONS:
Device: ELISIO dialyzer — 3 x week dialysis using ELISIO dialyzer for 12 weeks
  Other Names: ELISIOTM-H dialyzer
Device: Fresenius FX100 dialyzer

SUMMARY:
Today, haemodialysis is a recognized standard treatment for patients with chronic kidney disease stage 5. During the haemodialysis treatment session, blood passes from the patient through the extracorporeal circuit and is then returned. The dialyzer represents the greatest surface are of the extracorporeal circuit, as dialysis treatment is essentially based on the removal of small molecular weight solutes down along a concentration gradient, and this depends upon surface area. The ELISIO-H dialyzer differs in design to our current standard dialyzer, the FX100, by having fibers of a greater internal diameter, which potentially allows more internal haemofiltration, leading to an improved clearance of larger molecular weight solutes. It is now thought that these so called "middle molecular weight" solutes are more important in contributing to the clinical condition termed azotaemia, rather than smaller solutes such as urea.

The investigators therefore wish to study the clearance of middle sized molecules between the different dialyzers.

DETAILED DESCRIPTION:
Stable chronic kidney dialysis patients, currently dialyzing on the main Royal Free hospital dialysis unit will be asked to participate in the study. It is aimed to recruit 15 patients currently dialysing using the Fresenius FX100 dialyzer, who have used Fresenius polysulphone membranes for > 3 months.

During a mid week dialysis session, dialysis adequacy will be assessed by on line clearance, and samples of both blood and dialysate taken to assess, both clearances and bio-compatibility.

Thereafter patients would be switched to dialyse using the ELISIOTM-H dialyzer, but continue with the same dialysis prescription, and after 3 months, measurements repeated

Assessments Primary Clearances : on-line Kt/V, dual pool Kt/V, phosphate, b2microglobulin, cystatin C Secondary Serum :isoprostane generation complement activation platelet activation - coagulation activation - thrombophilic markers - Other Anticoagulation requirements & clotted circuits erythropoietin requirements, phosphate control therapy CRP

ELIGIBILITY:
Inclusion Criteria:

* 15 adult patients currently dialysing using the Fresenius FX100 dialyzer, who have used Fresenius polysulphone membranes for > 3 months, who are stable and able to provide informed consent.

Exclusion Criteria:

* using other dialyzers, unable to provide informed consent, unstable on dialysis or have problematical vascular access

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
solute clearances | 9 months

SECONDARY OUTCOMES:
erythropoietin requirements | 9 months
effect on inflammatory markers | 9 months
clotting potential | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: andrew davenport, md, Principal Investigator — center for nephrology, University college Hospital medical School
Locations (1):
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Vernon K, Peasegood J, Riddell A, Davenport A. Dialyzers designed to increase internal filtration do not result in significantly increased platelet activation and thrombin generation. Nephron Clin Pract. 2011;117(4):c403-8. doi: 10.1159/000319884. Epub 2010 Nov 12. PMID 21071966